CLINICAL TRIAL: NCT04890769
Title: Post Market Clinical Follow-up (PMCF) Study for DryMax Sensor
Brief Title: Clinical Study of Moisture Sensor Dressing Used for Exuding Wounds
Status: Terminated | Type: Observational
Why Stopped: The study is terminated by the sponsor due to poor participant recruitment and due to limited opportunity to achieve commercial gain.
Sponsor: Fredrik Iredahl (Other)
Collaborators: Primary Health Care Center, Department of Health Medicine and Caring Sciences, Linköping University, Linköping, Sweden (Unknown)
Responsible Party: Sponsor-Investigator, Fredrik Iredahl, Principal Investigator, Vårdcentralen Åby
Organization: Vårdcentralen Åby (Other)
Other Study IDs: 0007-P--047
Record Dates: First submitted 2021-04-26; First posted 2021-05-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Exuding Wounds; Ulcer, Leg; Wound
MeSH Terms: conditions — Leg Ulcer; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Patients with exuding wounds
  Interventions: Device: Moisture sensor wound dressing

INTERVENTIONS:
Device: Moisture sensor wound dressing — Clinical procedure for change of wound dressing
  Other Names: DryMax Sensor

SUMMARY:
Observational prospective study of the clinical use of a wound dressing with a moisture sensor for use on exuding wounds.

DETAILED DESCRIPTION:
The PMCF study will be performed as a prospective and open study of a wound dressing with a moisture sensor on exuding wounds.

Using DryMax Sensor and the display indication - advisory only - might influence the clinician's workflow and the patient's engagement in their care. The PMCF study aims to study the use of the sensor in the clinical procedure of dressing changes in one or more healthcare settings. To study how the new product is received, and how it is used in the workflow, related to its clinical performance.

Furthermore, the aim is to gather safety-related clinical data for common harms within exudate management.

ELIGIBILITY:
Inclusion Criteria:

* male or female, ≥18 years
* presence of an exuding wound, according to the clinician's assessment
* the wound is deemed suitable for treatment with DryMax Sensor
* an appropriate dressing size is available to be used according to the size of the wound
* the participant has given a written informed consent to participate in the study.

Exclusion Criteria:

* known pregnancy at the inclusion visit
* known or suspected hypersensitivity to the DryMax Sensor or its components
* mental inability, reluctance or language difficulties that cause difficulties in understanding the meaning of participating in the study
* ongoing treatment with systemic antibiotics
* illness or treatment of an indication other than the wound and which, according to the study personnel, can affect the wound treatment, the study, and/or the dressing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from primary health care
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Questionnaire regarding workflow of the clinical procedure for dressing change | Enrollment to study completion (4 weeks)
  Yes/no questions and questions with multiple choices
Questionnaire regarding the satisfaction using the device | Through study completion, up to 4 weeks
  Scale 1-5 where 1= low, 5 = good
Registration of device deficiencies | Enrollment to study completion (4 weeks)
  Type of device deficiency
Registration of device deficiencies | Enrollment to study completion (4 weeks)
  Severity scale 1-3, 1=low, 3=high

SECONDARY OUTCOMES:
Number of days between visits | Enrollment to study completion (4 weeks)
  Dressing change frequency
Weight of dressing after use using a balance | Enrollment to study completion (4 weeks)
  Utilisation of dressings capacity
Registration of time for display activation | Enrollment to study completion (4 weeks)
  Time for display activation - hours since application [h]
Questionnaire regarding leakage, strike-through, exudate viscosity | Enrollment to study completion (4 weeks)
  Yes/no questions and questions with multiple choices
Questionnaire regarding wound status | Enrollment to study completion (4 weeks)
  Questions with multiple choices
Measurement of wound size with a ruler | Enrollment to study completion (4 weeks)
  Wound size progression

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Iredahl, MD. PhD., Principal Investigator — Linkoeping University
Locations (1):
- Primary Health Care Center in Österlötland, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No
Data will be analyzed and published on a group level.